CLINICAL TRIAL: NCT02730650
Title: Assessing Outcomes for Platelet Rich Therapy for Facial Rejuvenation Using the FACE-Q Questionnaire
Brief Title: Platelet Rich Therapy for Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-00406
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Facial Rejuvenation
Keywords: FACE-Q; Platelet Rich Therapy; PRT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Platelet Rich Therapy (Experimental): Each subject will receive six injections of Platelet Rich Plasma (PRP) at designated points on each side of their face (twelve total). Injection points are spaced evenly across the inferior border of the cheek and mid-cheek, and are consistent on each patient. Patients will receive a post-injection phone call within 48 hours of the procedure. Photographs will be taken at two time points as part of the research to serve as a point of comparison before and after platelet rich plasma. Patients will receive the Global Aesthetic Improvement Scale amd tje Face-Q Questionnaire 1 month post-op
  Interventions: Other: Platelet Rich Therapy (PRT)

INTERVENTIONS:
Other: Platelet Rich Therapy (PRT) — Platelet Rich Therapy (PRT) involves injection of patient's own platelets and fibrin.Topical anesthetic will be applied to the face for a period of fifteen minutes prior to the injection. For PRP preparation, 8 cc of blood will be collected from each patient just before each procedure. Approximately 0.3-0.4 cc of PRP will be injected into each standardized injection point in a superficial manner. The injections points are 6 points on each side of the face along the inferior border of cheek and mid-cheek (12 total). The PRP injection will be followed by 10-15 minutes of icing.

SUMMARY:
This study will be a prospective study of patients who undergo platelet-rich therapy (PRT) for facial rejuvenation at NYU Langone Medical Center. PRT has been increasingly used for wound healing, fat grafting, hemostasis as well as facial enhancement. PRT involves injection of patient's own platelets and fibrin, and has evolved as a less invasive technique for facial rejuvenation compared to more traditional techniques. Through the use of pre and post treatment photos, in addition to the FACE-Q Questionnaire and a clinician assessment, it is our hope that we will confirm the rejuvenating capabilities of PRT.

DETAILED DESCRIPTION:
To assess patient-reported satisfaction of using platelet rich therapy for facial rejuvenation using a validated questionnaire (the FACE-Q scale). This is a prospective study of patients who will undergo platelet-rich therapy for facial rejuvenation at NYU Langone Medical Center. Platelet rich therapy (PRT) has been increasingly used for wound healing, fat grafting, hemostasis as well as facial enhancement. PRT involves injection of patient's own platelets and fibrin, and has evolved as a less invasive technique for facial rejuvenation compared to more traditional techniques. However, while platelet rich therapy for facial enrichment continues to gain popularity; little evidence exists to support its use in the current literature. Therefore, this study sets out to determine patient satisfaction as well as quality of life following PRT for facial rejuvenation. PRT has been previously used successfully in facial plastic surgery and is being offered as an option as part of standard of care for facial rejuvenation (Sclafani).

Subjects will be identified by the principal investigator as they present to the office for facial rejuvenation and are interested in an alternative to soft tissue fillers. All such patients will be given PRT as an alternative option for facial rejuvenation and any patient who agrees to this therapy will be enrolled in the study. Subject enrollment will continue until a total of 30 subjects are recruited.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Ages 21 - 80
* Patients of all racial and ethnic origins
* Patients of Dr. Hazen undergoing facial rejuvenation

Exclusion Criteria:

* Patients undergoing facial rejuvenation using other methods including botox injections, chemical peels, face lifts and others.
* Patients using blood thinners that cannot be stopped
* Patients who have used aspirin within a week of the procedure date

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction as measured by the FACE-Q scale | 1 Month Post-Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexes Hazen, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States